CLINICAL TRIAL: NCT05994807
Title: A Phase 1, Single-Center, Open-Label, 2-Cohort, Fixed-Sequence, Drug-Drug Interaction Study to Assess the Pharmacokinetics of DC-806 When Orally Administered Alone, When Coadministered With Itraconazole, and When Coadministered With Carbamazepine in Healthy Adult Participants
Brief Title: A Drug-Drug Interaction Study to Assess the Pharmacokinetics of DC-806 When Orally Administered Alone, When Coadministered With Itraconazole, and When Coadministered With Carbamazepine in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DICE Therapeutics, Inc., a wholly owned subsidiary of Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DCE806103
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Healthy Volunteers
Keywords: DC-806; Drug-Drug Interaction; Itraconazole; Carbamazepine
MeSH Terms: interventions — Itraconazole; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Participants in Cohort 1 will receive DC-806 single dose on Day 1, and the second dose of DC-806 along with itraconazole after the wash-out period.
  Interventions: Drug: DC-806; Drug: Itraconazole
- Cohort 2 (Experimental): Participants in Cohort 2 will receive DC-806 single dose on Day 1, and the second dose of DC-806 along with carbamazepine after the wash-out period.
  Interventions: Drug: DC-806; Drug: Carbamazepine

INTERVENTIONS:
Drug: DC-806 — Oral tablets
Drug: Itraconazole — Oral capsules
  Arms: Cohort 1
Drug: Carbamazepine — Oral tablets
  Arms: Cohort 2

SUMMARY:
The primary objective of this study is to assess the effect of a cytochrome P450 3A4 (CYP3A4) inhibitor (itraconazole) and CYP3A4 inducer (carbamazepine) on the single dose pharmacokinetics (PK) of DC-806 coadministered with itraconazole or carbamazepine in healthy male and female participants.

ELIGIBILITY:
Inclusion Criteria:

1. Sex : male or female; females must be of non-childbearing potential, or postmenopausal.
2. Age : 18 to 55 years, inclusive, at screening.
3. Body mass index (BMI) : 18.0 to 32.0 kg/m^2, inclusive, at screening.
4. Weight : ≥50 kg, inclusive, at screening.
5. Status : healthy participants. Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the investigator, active, or chronic disease.
6. Male participants and female participants of childbearing potential must agree to use protocol specified methods of contraception and comply with pregnancy precautions as described in the protocol.
7. All prescribed medication must have been stopped at least 14 days prior to admission to the clinical site.
8. All over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (e.g., St. John's wort) must have been stopped at least 7 days (or 5 half-lives for certain medications, whichever is longer) prior to admission to the clinical site. Occasional use of acetaminophen/paracetamol (e.g., up to 2 grams per day) is permitted during this period and throughout the study.
9. Ability and willingness to abstain from alcohol-, caffeine-, and methylxanthine-containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to admission to the clinical site and during confinement at the clinical site.
10. Willingness to abstain from any strenuous physical exercise from 96 hours (4 days) prior to admission and during confinement at the clinical site.
11. Good physical and mental health on the basis of medical history, physical examination, clinical laboratory assessments, 12-lead electrocardiogram (ECG), Columbia-Suicide Severity Rating Scale (C-SSRS) (Cohort 2 only) and vital signs, as judged by the Investigator.
12. Willing and able to sign the informed consent form (ICF).

Exclusion Criteria:

1. Employee of ICON or the Sponsor.
2. History of relevant drug and/or food allergies, in the opinion of the Investigator.
3. Females who are currently breastfeeding.
4. Smoking more than 5 cigarettes, 1 cigar, or 1 pipe daily within 3 months prior to screening.
5. Unwilling or unable to abstain from tobacco products within the 48 hours (2 days) prior to admission and during confinement at the clinical site.
6. History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within 1 year prior to screening.
7. Positive drug and/or alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at screening or admission to the clinical site.
8. History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average. Alcohol consumption will be prohibited 48 hours prior to admission to the clinical facility and until discharge in the study period.
9. Positive screen for hepatitis B surface antigen, hepatitis C virus (HCV) antibodies, or human immunodeficiency virus (HIV) 1 and 2 antibodies.
10. Consumption of any nutrients known to modulate cytochrome P450 (CYP450) enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to the first administration of study drug and during the study (including washout period/clinic furlough until after discharge in the last study period).
11. Participation in a drug study within 30 days prior to study drug administration in the current study. Participation in 4 or more other drug studies in the 12 months prior to study drug administration in the current study.
12. History of donation of more than 450 mL of blood within 60 days prior to dosing in the clinical site or planned donation before 30 days has elapsed since intake of study drug.
13. Plasma or platelet donation within 7 days of dosing and through follow-up.
14. Significant and/or acute illness within 5 days prior to study drug administration that may impact safety assessments, in the opinion of the Investigator.
15. Unsuitable veins for infusion or blood sampling as determined by the Investigator or study staff.
16. Any other condition or prior therapy that, in the Investigator's opinion, would confound or interfere with the evaluation of safety, tolerability, or pharmacokinetics (PK) of the study drug, interfere with study compliance, or preclude informed consent.

    Cohort 2 Only:
17. Individuals who have Asian ancestry (including those who have one or more Asian grandparents).
18. Presence of active suicidal ideation or positive suicide behavior using the "Baseline/Screening" version of the C-SSRS and with either of the following criteria:

    * History of a suicide attempt within the 5 years prior to the Screening Visit. Participants with a history of a suicide attempt more than 5 years ago should be evaluated by a mental healthcare professional (e.g., locally licensed psychiatrist, psychologist, or master's level therapist) before enrolling into the study.
    * Suicidal ideation in the past month prior to the Screening Visit as indicated by a positive response ("Yes") to either Question 4 or 5 of the "Baseline/Screening" version of the C-SSRS.
19. History of epilepsy.
20. Leukopenia (white blood cell count <lower limit of normal [LLN]), neutropenia (neutrophil count <LLN), or thrombocytopenia (platelet count <LLN), at screening or admission (Day -1).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Cohort 1: Maximum Observed Plasma Concentrations (Cmax) of DC-806 | Day 1 to Day 11
Cohort 2: Cmax of DC-806 | Day 1 to Day 25
Cohort 1: Area Under the Plasma Concentration-time Curve Up to Time t (AUC0-t) of DC-806 | Day 1 to Day 11
Cohort 2: AUC0-t of DC-806 | Day 1 to Day 25
Cohort 1: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity (AUC0-inf) of DC-806 | Day 1 to Day 11
Cohort 2: AUC0-inf of DC-806 | Day 1 to Day 25

SECONDARY OUTCOMES:
Cohorts 1 and 2: Number of Participants who Experience an Adverse Event | Up to a maximum of 31 days

CONTACTS AND LOCATIONS:
Locations (1):
- ICON Phase I Clinic, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No